CLINICAL TRIAL: NCT04907344
Title: A Multicenter, Open, Randomized Controlled Study of Camrelizumab+ Nab-paclitaxel + Carboplatin Versus Nab-paclitaxel + Carboplatin as Neoadjuvant Therapy for Triple Negative Breast Cancer (TNBC)
Brief Title: Study of Camrelizumab Plus Chemotherapy as Neoadjuvant Therapy in Participants With Triple Negative Breast Cancer (TNBC)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Zhongsheng Tong, Director of Breast Oncology, Tianjin Medical University Cancer Institute and Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-BC-II-024
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — camrelizumab; 130-nm albumin-bound paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1: Camrelizumab + Chemotherapy (Experimental)
  Interventions: Drug: Camrelizumab; Drug: Nab-Paclitaxel; Drug: Carboplatin
- Part 2: Camrelizumab + Chemotherapy (Experimental)
  Interventions: Drug: Camrelizumab; Drug: Nab-Paclitaxel; Drug: Carboplatin
- Part 2: Chemotherapy (Active Comparator)
  Interventions: Drug: Nab-Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Camrelizumab — IV infusion
  Arms: Part 1: Camrelizumab + Chemotherapy; Part 2: Camrelizumab + Chemotherapy
Drug: Nab-Paclitaxel — IV infusion
Drug: Carboplatin — IV infusion

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Camrelizumab in Combination With Nab-Paclitaxel and carboplatin as Neoadjuvant Therapy in Participants With Triple Negative Breast Cancer (TNBC).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed breast cancer;
* 18-75 Years, female;
* ECOG Performance Status of 0-1;
* Life expectancy is not less than 3 months;
* Histologically documented TNBC (negative human epidermal growth factor receptor 2 [HER2], estrogen receptor [ER], and progesterone receptor [PgR] status);
* Tumor stage: II-III;
* At least one measurable lesion according to RECIST 1.1;
* Adequate hematologic and organ function.;
* Must be willing to use an adequate method of contraception for the course of the study.

Exclusion Criteria:

* Stage Ⅳ (metastatic) breast cancer or bilateral breast cancer;
* Inflammatory breast cancer;
* Has received prior any anti-tumor therapy within the past 12 months prior to signing informed consent, including chemotherapy, targeted therapy, radiation therapy, immunotherapy, biotherapy and TACE;
* Has received prior therapy with an anti-programmed cell death protein 1 (anti-PD-1), anti-programmed death - ligand 1 (anti-PD-L1), or anti-PD-L2 agent or with an agent directed to another co-inhibitory T-cell receptor (e.g., cytotoxic T-lymphocyte-associated antigen-4 [CTLA-4];
* Has a history of invasive malignancy ≤5 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer;
* Major surgical procedure within 4 weeks prior to initiation of study treatment;
* Active or history of autoimmune disease or immune deficiency diseases except history of autoimmune-related hypothyroidism, controlled Type 1 diabetes mellitus;
* Has a history of (non-infectious) pneumonitis, interstitial lung disease or uncontrollable systematicness diseases;
* Administration of a live attenuated vaccine within 28 days prior to initiation of study treatment or anticipation of need for such a vaccine during the study;
* Has a known history of Human Immunodeficiency Virus (HIV);
* Has known active Hepatitis B, Hepatitis C or Autoimmune hepatitis;
* Severe infections within 4 weeks prior to initiation of study treatment, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia;
* Has active infection (CTCAE≥2) needed the treatment of antibiotic within 2 weeks prior to initiation of study treatment;
* Has evidence of active tuberculosis within 1year prior to initiation of study treatment;
* Prior allogeneic stem cell or solid organ transplantation;
* Pre-existing motor or sensory neuropathy of a severity≥grade 2;
* Has significant cardiovascular disease;
* Has a known hypersensitivity to the components of the study treatment or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins;
* Female patients during pregnancy and lactation, fertile women with positive baseline pregnancy tests or women of childbearing age who are unwilling to take effective contraceptive measures throughout the trial;
* History of neurological or psychiatric disorders, including epilepsy or dementia;
* Any other situation evaluated by researchers.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2021-06-15 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
pCR rate using the definition of ypT0/Tis ypN0 (i.e., no invasive residual in breast or nodes; noninvasive breast residuals allowed) at the time of definitive surgery | Up to approximately 24 weeks
  pCR rate (ypT0/Tis ypN0) is defined as the percentage of participants without residual invasive tumor on hematoxylin and eosin evaluation of breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy by current AJCC staging criteria assessed by the local pathologist at the time of definitive surgery in all participants.

SECONDARY OUTCOMES:
pCR rate using the definition of ypT0/Tis (i.e., absence of invasive cancer in the breast irrespective of ductal carcinoma in situ or nodal involvement) at the time of definitive surgery | Up to approximately 24 weeks
  pCR rate (ypT0/Tis) is defined as the percentage of participants without invasive cancer in the breast irrespective of ductal carcinoma in situ or nodal involvement following completion of neoadjuvant systemic therapy by current AJCC staging criteria assessed by the local pathologist at the time of definitive surgery in all participants
Objective Response Rate (ORR) | Up to approximately 24 weeks
  ORR was defined as percentage of participants with best (confirmed) overall response (BOR) of either CR or PR. ORR was assessed by the investigator according to RECIST version 1.1 and is based on BOR, which is defined as best response recorded from start of study treatment until definitive surgery or disease progression.
Event-Free Survival (EFS) | Up to approximately 5 years
  EFS is defined as the time from start of study treatment to any of the following events: progression of disease that precludes surgery, local or distant recurrence, second primary malignancy (breast or other cancers) or death due to any cause.
Invasive Disease-Free Survival (iDFS) | Up to approximately 5 years
  iDFS events are defined as follows: (1)Ipsilateral invasive breast tumor recurrence. (2) Ipsilateral local-regional invasive breast cancer recurrence. (3) Ipsilateral second primary invasive breast cancer. (4) Contralateral invasive breast cancer. (5) Distant recurrence. (6) Death attributable to any cause.
Overall survival (OS) | Up to approximately 5 years
  OS is defined as the time from randomization to death due to any cause. Participants without documented death at the time of the analysis will be censored at the date of the last follow-up.
Adverse events (AEs) | Up to approximately 35 weeks
  AEs were graded according to the National Cancer Institute's Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0.
  In general, AEs are graded according to the following: Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE.
  The type, grade and frequency of AEs will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Zhongsheng Tong, MD, Principal Investigator — Breast Oncology, Tianjin Medical University Cancer Institute and Hospital; Xuchen Cao, MD, Principal Investigator — Breast Cancer Department I, Tianjin Medical University Cancer Institute and Hospital
Locations (2):
- China (2):
  - Breast Cancer Department I, Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Breast Oncology, Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality